CLINICAL TRIAL: NCT01963650
Title: Natural History Study of Children With Metachromatic Leukodystrophy
Status: Terminated | Type: Observational
Why Stopped: Enrollment issues
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-MLD-092
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Lipid Metabolism Disorders; Metachromatic Leukodystrophy (MLD); Nervous System Diseases; Brain Diseases; Central Nervous System Diseases; Demyelinating Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Sphingolipidoses; Hereditary Central Nervous System Demyelinating Diseases; Metabolic Inborn Brain Diseases; Lysosomal Storage Diseases; Metabolic Diseases; Sulfatidosis
MeSH Terms: conditions — Lipid Metabolism Disorders; Leukodystrophy, Metachromatic; Nervous System Diseases; Brain Diseases; Central Nervous System Diseases; Demyelinating Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Sphingolipidoses; Hereditary Central Nervous System Demyelinating Diseases; Brain Diseases, Metabolic, Inborn; Lysosomal Storage Diseases; Metabolic Diseases; Sulfatidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample for genotype testing is collected and any remaining sample is retained for follow up or repeat testing. The sample is not retained for unspecified additional testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The purpose of this study is evaluate the natural course of disease progression related to gross motor function in children with metachromatic leukodystrophy (MLD).

DETAILED DESCRIPTION:
Metachromatic leukodystrophy (MLD) is an inherited, autosomal recessive disorder of lipid metabolism characterized by deficient activity of the lysosomal enzyme, arylsulfatase A (ASA). MLD is a rare genetic disease that occurs in most parts of the world. The estimated overall incidence of the disease in the western world is approximately 1 in 100,000 live births.

This study is a multicenter, observational, longitudinal study that plans to enroll up to 30 patients with onset of MLD-related signs and symptoms prior to 30 months of age and who are less than 12 years of age. Patients will participate in this study for approximately 114 weeks (Screening through Follow-up) and will be assessed at defined intervals for disease status.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of MLD by both:

   * arylsulfatase A (ASA) deficiency by assay in leukocytes AND
   * elevated sulfatide in urine
2. Appearance of the first symptoms of disease at or before 30 months of age.
3. A GMFM-88 total (percent) score greater than or equal to 40 at the screening examination.
4. The patient is less than 12 years of age at the time of enrollment.
5. The patient and his/her parent or legally authorized representative(s) must have the ability to comply with the clinical protocol.
6. Patient's parent or legally authorized representative(s) must provide written informed consent prior to performing any study-related activities. Study-related activities are any procedures that would not have been performed during normal management of the patient.

Exclusion Criteria:

1. History of hematopoietic stem cell transplantation.
2. The patient has any known or suspected hypersensitivity to agents used for anesthesia or is thought to be at an unacceptably high risk for associated potential complications of airway compromise or other conditions.
3. Any other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study.
4. The patient is enrolled in another clinical study that involves the use of any investigational product (drug or device) within 30 days prior to study enrollment or at any time during the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll up to 30 male or female children (<12 years of age) with a confirmed MLD diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the change from baseline in motor function using the GMFM-88 total (percent) score. | Week 0 to Week 104

SECONDARY OUTCOMES:
The change from baseline in ability to swallow as assessed by the Functional Endoscopic Evaluation of Swallowing. | Week 0 to Week 104
The change from baseline in nerve conduction as measured by the electroneurography. | Week 0 to Week 104
The change from baseline in the adaptive behavior composite standard score as measured by the Vineland Adaptive Behavior Scales. | Week 0 to Week 104
The change from baseline in domain-specific Caregiver Observed MLD Functioning and Outcomes Reporting Tool. | Week 0 to Week 104
The change from baseline in cognitive function using the Mullen Scales of Early Learning. | Week 0 to Week 104
Reporting of any study procedure-related nonserious AEs and/or any SAEs | Week 0 to Week 114

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (4):
  - Harbor UCLA Pediatrics, Torrance, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital Of Pittsburgh, Pittsburgh, Pennsylvania
- Hospital Universitario Austral, Pilar, Argentina
- Universitair Ziekenhuis Antwerpen (UZA) (University Hospital Antwerpen), Edegem, Belgium
- Hospital de Cllnicas de Porto Alegre (HCPA) / UFRGS, Porto Alegre, Brazil
- Montreal Children's Hospital, Westmount, Canada
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- Hôpital De Bicêtre, Le Kremlin-Bicêtre, France
- Univesitatsklinikum Tubingen Klinik fur Kinder und Jugendmedizin, Tübingen, Germany
- Japan (2):
  - Faculty Of Medicine, Osaka University Graduate School Of Medicine, Osaka
  - The Jikei University School Of Medicine - Institute Of Dna Medicine, Tokyo
- Hacettepe Universitesi Tip Fakultesi Onkoloji Hastanesi, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fce4db2bf003ab467b3